CLINICAL TRIAL: NCT02864472
Title: Comparison of Early Intervention of PDT Combination With Ranibizumab vs. Ranibizumab Monotherapy in Persistent PCV Patients With Initial Loading Dose
Brief Title: Comparison of PDT Combination With Ranibizumab vs. Ranibizumab Monotherapy in Persistent PCV With Initial Loading Dose
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: CRFB002AKR16T
Record Dates: First submitted 2016-08-04; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — 1-phenyl-3,3-dimethyltriazene; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- combination Tx (Other): combination Tx(vPDT +ranibizumab) (M0) + ranibizumab PRN (M3-6)
  Interventions: Procedure: PDT; Drug: ranibizumab PRN
- mono Tx (Other): Ranibizumab (at 4 weeks interval) *3 (M0-2) + ranibizumab PRN (M3-6)
  Interventions: Drug: Ranibizumab; Drug: ranibizumab PRN

INTERVENTIONS:
Procedure: PDT — PDT and ranibizumab
  Arms: combination Tx
Drug: Ranibizumab — Ranibizumab
  Other Names: Lucentis
  Arms: mono Tx
Drug: ranibizumab PRN — ranibizumab PRN
  Other Names: Lucentis

SUMMARY:
The aim of this study is to compare the efficacy of early intervention of PDT combination compared with consecutive monthly treatment of intravitreal ranibizumab injections in PCV patients showing insufficient response with initial loading dose.

DETAILED DESCRIPTION:
PCV is generally recognized as a subtype of wet AMD characterized by the presence of aneurysmal orange-red polypoidal lesions with or without branching vascular network (BVN) in the choroidal vasculature as observed on indocyanine angiography (ICGA), representing 13% to 54.7% of newly diagnosed patients with neovascular AMD. Fifty percent of PCV had persistent leakage or recurrent bleeding with poor visual outcome, if left untreated.

And in the EVEREST study has shown that synergistic effects of anti-VEGF and vPDT combination: vPDT strongly regress polyp and anti-VEGF control to up-regulation of VEGF induced by vPDT compared to ranibizumab monotherapy in newly diagnosed PCV patients. Additionally, combination offers an opportunity for individualized treatment with potentially fewer treatments and less costs.

Therefore, the aim of this study is to compare the efficacy of early intervention of PDT combination compared with consecutive monthly treatment of intravitreal ranibizumab injections in PCV patients showing insufficient response with initial loading dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal to or older than 50 years
2. Insufficient responder to ranibizumab Tx
3. ICGA-confirmed PCV
4. BCVA letter score of 73 to 24 using Early Treatment of Diabetic Retinopathy Study charts
5. Ability to provide written informed consent and comply with study assessments for the full duration of the study

Exclusion Criteria:

1. Prior treatment with other anti-VEGF treatments in the study eye.
2. Prior treatment with other anti-VEGF treatments within 3 months prior to Visit 1 in the non-study eye.
3. Prior treatment with verteporfin within 6 months prior to Visit 1 in the study eye.
4. Prior treatment with verteporfin within 7 days prior to Visit 1 in the non-study eye.
5. Previous subfoveal focal laser photocoagulation involving the foveal center in the study eye
6. Previous submacular surgery in the study eye
7. A history of angioid streaks, presumed ocular histoplasmosis syndrome, or pathologic myopia
8. Experienced RPE tear, retinal detachment, macular hole, or uncontrolled glaucoma
9. Previous participation in a clinical trial involving anti-angiogenic drugs
10. Intraocular surgery: 2 months before Visit 1 in the study eye.
11. Previous participation in any studies of investigational drugs
12. Administration of periocular, intravitreal, or systemic corticosteroid in the previous 3 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-06 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change in central retinal thickness | after 6month
  Change in central retinal thickness measured by OCT

SECONDARY OUTCOMES:
Change of ETDRS BCVA | after 6month
  Change of ETDRS BCVA from baseline to 26 weeks and time course of it

CONTACTS AND LOCATIONS:
Overall Officials: Jangwon Heo, MD, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] 1. Wong RLM et al. J Ophthalmol Vis Res 2013;8:359-71. 2. Koh A et al. Retina 2013;33:686-716 3. Nakashizuka H et al. Invest Ophthalmol Vis Sci 2008;49:4729-37 4. Gomi F, Tano Y Curr Opin Ophthalmol 2008;19:208-12 5. Honda S et al. Ophthalmologica 2014;231:59-74 6. Maruko E et al. Am J Ophthalmol 2007;144:15-22 7. Byeon S et al. Jpn J Ophthalmol 2008;52:57-62 8. Uyama M et al. Am J Ophthalmol 2002;133:639-48